CLINICAL TRIAL: NCT03056690
Title: A Phase 2a, Randomized, Double-Blind Placebo-controlled, Parallel-group Study to Assess the Analgesic Efficacy and Safety of ASP0819 in Patients With Fibromyalgia
Brief Title: A Study to Assess the Analgesic Efficacy and Safety of ASP0819 in Patients With Fibromyalgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0819-CL-0201
Record Dates: First submitted 2017-02-15; First posted 2017-02-17 (Actual); Results first posted 2021-03-03 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Fibromyalgia
Keywords: ASP0819; Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ASP0819 (Experimental): Participants received ASP019 15 mg capsules, orally, once daily in the morning, with or without food for 8 weeks.
  Interventions: Drug: ASP0819
- Placebo (Placebo Comparator): Participants received ASP019 matching placebo capsules, orally, once daily in the morning, with or without food for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP0819 — Oral capsule
  Arms: ASP0819
Drug: Placebo — Oral capsule
  Arms: Placebo

SUMMARY:
This study assessed analgesic efficacy of ASP0819 relative to placebo as well as the safety and tolerability.

This study assessed treatment differences in physical function as well as the improvements in overall subject status (e.g., fibromyalgia symptoms and global functioning) of ASP0819 relative to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body mass index (BMI) ≤ 45 kg/m2.
* Female subject must either:

  * Be of nonchildbearing potential: postmenopausal (defined as at least 1 year without any menses) prior to Screening, or documented surgically sterile (e.g., hysterectomy, bilateral salpingectomy, bilateral oophorectomy).
  * Or, if of childbearing potential: agree not to try to become pregnant during the study and for 28 days after the final study drug administration, have a negative blood pregnancy test at Screening and negative urine test on Day 1, and if heterosexually active, agree to consistently use 1 form of highly effective birth control starting at Screening and throughout the study period and for 28 days after the final study drug administration.
* Female subject must agree not to breastfeed at Screening and throughout the study period, and for 28 days after the final study drug administration.
* Female subject must not donate ova starting at Screening, throughout the study period, and for 28 days after the final study drug administration
* Male subject must not donate sperm starting at Screening and throughout the study period, and for 28 days after the final study drug administration.
* Male subject with a partner of child-bearing potential, or a pregnant or breastfeeding partner(s) must agree to remain abstinent or use a condom throughout the study period and for 28 days after the final study drug administration.
* Subject meets the American College of Rheumatology (ACR) 1990 fibromyalgia diagnostic criteria at Screening:

  * Widespread pain for at least 3 months, defined as the presence of all of the following: pain on right and left sides of the body, pain above and below the waist, and pain in the axial skeleton (cervical spine or anterior chest or thoracic spine or low back) must be present.
  * Pain in at least 11 of 18 tender point sites on digital palpation. Digital palpation should be performed with an approximate force of 4 kg.
* Subject meets the ACR 2010 fibromyalgia diagnostic criteria at Screening:

  * Widespread pain index (WPI) ≥ 7 and Symptom severity (SS) scale score ≥ 5 or WPI 3-6 and SS scale score ≥ 9.
  * Symptoms have been present at a similar level for at least 3 months.
  * The subject does not have a disorder that would otherwise explain the pain.
* Subject has a pain score ≥ 4 on the revised fibromyalgia impact questionnaire revised (FIQR) pain item at Screening.
* Subject is compliant with daily pain recordings during the Baseline Diary Run-In period, as defined by the completion of a minimum of 5 of 7 daily average pain ratings and agrees to complete daily diaries throughout the duration of the study.
* Subject has a mean daily average pain score ≥ 4 and ≤ 9 on an 11-point 0 to 10 NRS as recorded in the subject e-diary during the Baseline Diary Run-In period, and meeting pre-specified criteria for daily average pain scores.
* Subject agrees to use only acetaminophen as rescue medication for fibromyalgia pain throughout the course of the trial (up to 1000 mg per dose and not to exceed 3000 mg/day).
* Subject agrees not to initiate or change any non-pharmacologic interventions (including normal daily exercise routines, chiropractic care, physical therapy, psychotherapy, and massage therapy) during the course of the study. Non-pharmacologic interventions must be stable for a minimum of 30 days prior to Screening. The subject agrees to maintain usual level of activity for the duration of the study.
* Subject is capable of completing study assessments and procedures.
* Subject agrees not to participate in another interventional study from Screening through the End of Study (EOS) visit.

Exclusion Criteria:

* Subject has received an investigational therapy within 28 days or 5 half-lives, whichever is longer, prior to Screening.
* Subject has had no meaningful improvement, from 2 or more prior treatments (commercially available) for fibromyalgia (in at least 2 pharmacologic classes).
* Subject has had known hypersensitivity or intolerance to the use of acetaminophen or associated formulation components; known hypersensitivity to the formulation components of ASP0819.
* Subject has pain due to diabetic peripheral neuropathy, post-herpetic neuralgia, traumatic injury, prior surgery, complex regional pain syndrome, or other source of pain that would confound or interfere with the assessment of the subject's fibromyalgia pain or require excluded therapies during the subject's study participation.
* Subject has infectious or inflammatory arthritis (e.g., rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis and gout), autoimmune disease (e.g., systemic lupus erythematosus), or other widespread rheumatic disease other than fibromyalgia.
* Subject has a current, untreated moderate or severe major depressive disorder as assessed by the Mini-International Neuropsychiatric Interview (M.I.N.I.). Subject with current, treated major depressive disorder can be included provided that it is without clinically significant changes in symptoms while on the same dose of a protocol allowed antidepressant for greater than 60 days prior to Screening.
* Subject has initiated any non-pharmacologic interventions for the treatment of fibromyalgia or depression within 30 days prior to Screening or during the Screening period.
* Subject has a history of any psychotic and/or bipolar disorder as assessed by the M.I.N.I.
* Subject has a Hospital Anxiety and Depression Scale (HADS) score > 14 on the Depression subscale at Screening or at the time of Visit 3 (Randomization).
* Subject has a history of suicide attempt or suicidal behavior within the last 12 months, or has suicidal ideation within the last 12 months (a response of "yes" to questions 4 or 5 on the suicidal ideation portion of the Columbia-Suicide Severity Rating Scale (C-SSRS)), or who is at significant risk to commit suicide at the time of Visit 3 (Randomization).
* Subject has clinically significant abnormalities in clinical chemistry, hematology, or urinalysis, or a serum creatinine > 1.5 times the Upper limit of normal (ULN) at Screening. These assessments may be repeated once, after a reasonable time period (but within the Screening period).
* Subject has aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥ 1.5 times the upper limit of the reference range at Screening. These assessments may be repeated once, after a reasonable time period (but within the Screening period).
* Subject has a positive test for hepatitis B surface antigen (HBsAg), hepatitis A virus antibodies (immunoglobulin M) (anti-HAV [IgM]) or hepatitis C virus antibodies (anti-HCV) at Screening or has history of a positive test for human immunodeficiency virus type 1(HIV-1) and/or type 2 (HIV-2).
* Subject has a resting systolic blood pressure (SBP) > 180 mmHg or < 90 mmHg, and/or a sitting diastolic blood pressure (DBP) > 100 mmHg at Screening. These assessments may be repeated once, after a reasonable time period (but within the Screening period).
* Subject has a clinically significant abnormality on 12-lead Electrocardiogram (ECG) at Screening or Visit 3 (Randomization). If the ECG is abnormal, an additional ECG can be carried out. If this also gives an abnormal result, the subject must be excluded.
* Subject has a history of myocardial infarction (within 6 months of Screening), unexplained syncope, cardiac arrest, unexplained cardiac arrhythmias or torsade de pointes, structural heart disease or a family history of Long time from electrocardiogram Q wave to the end of the T wave (QT) Syndrome.
* Subject has evidence of any clinically significant, uncontrolled cardiovascular, gastrointestinal, endocrinologic (low thyroid stimulating hormone [TSH], but euthyroid is allowed), hematologic, hepatic, immunologic, infectious, metabolic, urologic, pulmonary (including obstructive sleep apnea not controlled by a Continuous positive airway pressure (CPAP) device) neurologic, dermatologic, psychiatric, renal and/or other major disease (exclusive of fibromyalgia).
* Subject has planned surgery during the study participation.
* Subject has an active malignancy or a history of malignancy (except for treated nonmelanoma skin cancer) within 5 years of Screening.
* Subject has a positive drug or alcohol test at Screening, Baseline Diary Run-In or prior to Randomization. However, a positive test for tetrahydrocannabinol (THC) and/or opioids is allowed at the Screening visit, but must be confirmed negative prior to Baseline Diary Run-In and Randomization.
* Subject has a current or recent (within 12 months of Screening) history of a substance use disorder including cannabinoid and/or alcohol abuse disorder. Subject has used opioids for pain for more than 4 days during the week preceding the Screening visit.
* Subject is currently using protocol specified prohibited medications and is unable to wash-out.
* Subject has filed or is awaiting judgment on a disability claim or has any pending worker's compensation litigation or related monetary settlements.
* Subject is an employee of the Astellas Group, the Contract Research Organization (CRO) involved, or the investigator site personnel directly affiliated with this study and/or their immediate families (spouse, parent, child, or sibling, whether biological or legally adopted).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2018-02-27 (Actual); Study Completion 2018-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (24):
- United States (24):
  - Site US10025 - Achieve Clinical Research, LLC, Birmingham, Alabama
  - Site US10045 - TriWest Research Associates, El Cajon, California
  - Site US10039 - Superior Research LLC, Sacramento, California
  - Site US10003 - Artemis Inst For Clin Research, San Diego, California
  - Site US10048 - Diablo Clinical Research Inc, Walnut Creek, California
  - Site US10028 - Renstar Medical Research, Ocala, Florida
  - Site US10024 - Compass Research LLC, Orlando, Florida
  - Site US10012 - Palm Beach Research Center, West Palm Beach, Florida
  - Site US10056 - Atlanta Ctr for Med Research, Atlanta, Georgia
  - Site US10006 - Columbus Regional Research Ins, Columbus, Georgia
  - Site US10038 - Heartland Research Associates, Wichita, Kansas
  - Site US10055 - Central Kentucky Research Asc, Lexington, Kentucky
  - Site US10027 - BTC of New Bedford LLC, New Bedford, Massachusetts
  - Site US10018 - Altea Research Institute, Las Vegas, Nevada
  - Site US10010 - Upstate Clinical Research Asc, Williamsville, New York
  - Site US10032 - Peters Medical Research, High Point, North Carolina
  - Site US10031 - Wake Research Associates, Raleigh, North Carolina
  - Site US10019 - Lillestol Research LLC, Fargo, North Dakota
  - Site US10037 - Dept of Psychiatry and Neuro University of Cincinnati, Cincinnati, Ohio
  - Site US10059 - Hillcrest Clinical, Oklahoma City, Oklahoma
  - Site US10043 - Oregon Ctr for Clinical Invest, Portland, Oregon
  - Site US10023 - Oregon Ctr for Clinical Invest, Salem, Oregon
  - Site US10013 - Bateman Horne Center, Salt Lake City, Utah
  - Site US10005 - Charlottesville Med Research, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Arnold LM, Blauwet MB, Tracy K, Cai N, Walzer M, Blahunka P, Marek GJ. Efficacy and Safety of ASP0819 in Patients with Fibromyalgia: Results of a Proof-of-Concept, Randomized, Double-Blind, Placebo-Controlled Trial. J Pain Res. 2020 Dec 10;13:3355-3369. doi: 10.2147/JPR.S274562. eCollection 2020. PMID 33328761
- See also: Link to results on the Astellas Clinical Study Results website. — https://astellasclinicalstudyresults.com/study.aspx?ID=344

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male and female participants between 18 and 80 years of age with fibromyalgia were enrolled in this study.
Groups:
- Placebo: Participants received ASP0819 matching placebo capsules, orally, once daily in the morning, with or without food for 8 weeks.
- ASP0819 15mg: Participants received ASP0819 15 mg capsules, orally, once daily in the morning, with or without food for 8 weeks.
Period: Overall Study
Arm/Group | Placebo | ASP0819 15mg
Started | 95 | 91
Treated | 94 | 90
Completed | 81 | 75
Not Completed | 14 | 16
Not completed — Adverse Event | 3 | 2
Not completed — Lack of Efficacy | 1 | 2
Not completed — Lost to Follow-up | 3 | 2
Not completed — Protocol Violation | 2 | 2
Not completed — Withdrawal by Subject | 3 | 6
Not completed — Non-compliance with Study Drug | 1 | 0
Not completed — Miscellaneous | 1 | 2

BASELINE CHARACTERISTICS:
Population: All participants who were randomized to this study.
Groups:
- ASP0819 15 mg: Participants received ASP0819 15 mg capsules, orally, once daily in the morning, with or without food for 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | ASP0819 15 mg | Total
Number analyzed (Participants) | 95 | 91 | 186
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.9 (12.5) | 48.7 (12) | 49.3 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 89 | 179
  Male | 5 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 10 | 23
  Not Hispanic or Latino | 82 | 81 | 163
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 16 | 11 | 27
  White | 74 | 78 | 152
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Mean Daily Average Pain Score [Mean (Standard Deviation); unit: Units on a scale] — The mean daily average pain score is assessed by numerical rating scale (NRS). The NRS is a generic instrument for the assessment of pain, consisting of a single question that asks participants to record their daily average pain on an 11-point scale, where 0 anchors "no pain" and 10 "pain as bad as you can imagine". Mean daily average pain score was assessed over a 1 week baseline diary run-in period. Population: The full analysis set (FAS) consisted of all participants who were randomized and received at least 1 dose of study drug.
  Units on a scale
    number analyzed (Participants) | 94 | 90 | 184
    (all) | 6.32 (1.02) | 6.32 (1.01) | 6.32 (1.01)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 8 in Mean Daily Average Pain Score Assessed by NRS
Description: The change from baseline to Week 8 in mean daily average pain score is assessed by NRS. The NRS is a generic instrument for the assessment of pain, consisting of a single question that asks participants to record their daily average pain on an 11-point scale, where 0 anchors "no pain" and 10 "pain as bad as you can imagine". A negative change indicates a reduction/improvement from baseline (i.e. a favorable outcome).
Time Frame: Baseline and week 8
Population: FAS population
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | ASP0819 15 mg
Number analyzed (Participants) | 81 | 75
Units on a scale | -1.26 (0.18) | -1.60 (0.18)
Statistical Analysis 1: Comparison: Placebo vs ASP0819 15 mg; Test type: Superiority — Mixed model repeated measures (MMRM) analysis model is performed with change from baseline (Week 8) as response; treatment, center (pooled where necessary), time (week 8) and treatment*time as fixed effects, baseline and baseline*time as covariates; p = 0.086, MMRM; LSMean Difference = -0.34, 90% CI 2-sided [-0.76 to 0.07], Standard Error of Mean 0.25

2. Primary Outcome: Number of Participants With Adverse Events
Description: TEAE was defined as any AE which started, or worsened, after the first dose of study drug through 30 days after the last dose of study drug. AE was considered serious if: resulted in death, was life- threatening, resulted in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, resulted in congenital anomaly or birth defect, required inpatient hospitalization or led to prolongation of hospitalization, other medically important events.
Time Frame: From first dose of study drug until end of study (up to Day 85)
Population: The safety analysis set (SAF) consisted of all randomized participants who took at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Placebo | ASP0819 15 mg
Number analyzed (Participants) | 94 | 90
Participants
  Treatment emergent adverse event (TEAE) | 53 | 62
  Serious TEAE | 0 | 0

3. Primary Outcome: Number of Participants With Suicidal Ideation and Suicidal Behavior at Week 2
Description: C-SSRS was used for suicide assessment. Participants were asked detailed questions regarding suicidal ideation, behaviors, intensity of ideation, and attempts. Suicidal ideation: A "yes" answer to any one of the following five questions from suicidal ideation section on the C-SSRS. 1. Wish to be dead 2. Non-specific active suicidal thoughts 3. Active suicidal ideation with any methods (not plan) without intent to act 4. Active suicidal ideation with some intent to act, without specific plan 5. Active suicidal ideation with specific plan and intent. Suicidal behavior: "yes" answer to any one of the following five questions from suicidal behavior section on the C-SSRS. 6. Preparatory acts or behavior 7. Aborted attempt 8. Interrupted attempt 9. Actual attempt 10. Completed suicide.
Time Frame: Week 2
Population: SAF population with available data at specified time point.
Measure: Number; unit: Participants
Arm/Group | Placebo | ASP0819 15 mg
Number analyzed (Participants) | 89 | 90
Participants
  Week 2: Suicidal Ideation | 0 | 0
  Week 2: Suicidal Behavior | 0 | 0

4. Primary Outcome: Number of Participants With Suicidal Ideation and Suicidal Behavior at Week 4
Description: as for outcome 3
Time Frame: Week 4
Population: SAF population with available data at specified time point.
Measure: Number; unit: Participants
Arm/Group | Placebo | ASP0819 15 mg
Number analyzed (Participants) | 89 | 90
Participants
  Week 4: Suicidal Ideation | 0 | 0
  Week 4: Suicidal Behavior | 0 | 0

5. Primary Outcome: Number of Participants With Suicidal Ideation and Suicidal Behavior at Week 8
Description: as for outcome 3
Time Frame: Week 8
Population: SAF population with available data at specified time point.
Measure: Number; unit: Participants
Arm/Group | Placebo | ASP0819 15 mg
Number analyzed (Participants) | 79 | 74
Participants
  Week 8: Suicidal Ideation | 0 | 0
  Week 8: Suicidal Behavior | 0 | 0

6. Primary Outcome: Number of Participants With Suicidal Ideation and Suicidal Behavior at Week 10
Description: C-SSRS was used for suicide assessment. Participants were asked detailed questions regarding suicidal ideation, behaviors, intensity of ideation, and attempts. Suicidal ideation: A "yes" answer to any one of the following five questions from suicidal ideation section on the C-SSRS. 1. Wish to be dead 2. Non-specific active suicidal thoughts 3. Active suicidal ideation with any methods (not plan) without intent to act 4. Active suicidal ideation with some intent to act, without specific plan 5. Active suicidal ideation with specific plan and intent Suicidal behavior: "yes" answer to any one of the following five questions from suicidal behavior section on the C-SSRS. 6. Preparatory acts or behavior 7. Aborted attempt 8. Interrupted attempt 9. Actual attempt 10. Completed suicide.
Time Frame: Week 10
Population: SAF population with available data at specified time point.
Measure: Number; unit: Participants
Arm/Group | Placebo | ASP0819 15 mg
Number analyzed (Participants) | 88 | 85
Participants
  Week 10: Suicidal Ideation | 1 | 0
  Week 10: Suicidal Behavior | 0 | 0

7. Secondary Outcome: Percentage of Participants Achieving Greater Than or Equal to (≥)30 % Reduction From Baseline to Week 8 in Mean Daily Average Pain Score Assessed by NRS
Description: The mean daily average pain score is assessed by NRS. The NRS is a generic instrument for the assessment of pain, consisting of a single question that asks participants to record their daily average pain on an 11-point scale, where 0 anchors "no pain" and 10 "pain as bad as you can imagine".
Time Frame: Baseline and week 8
Population: FAS population with baseline observation carried forward (BOCF) imputation.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | ASP0819 15 mg
Number analyzed (Participants) | 94 | 90
Percentage of participants | 29.8 [22.1 to 38.5] | 30.0 [22.1 to 38.9]
Statistical Analysis 1: Comparison: Placebo vs ASP0819 15 mg; Test type: Superiority; p = 0.551, Fisher Exact; CI for each treatment group and the difference of the proportions is an exact unconditional confidence interval based on Santner-Snell approach; Difference = 0.2, 90% CI 2-sided [-11.9 to 12.5]

8. Secondary Outcome: Percentage of Participants Achieving ≥ 30 % Reduction From Baseline to End of Treatment (EOT) in Mean Daily Average Pain Score Assessed by NRS
Description: The mean daily average pain score is assessed by NRS.The NRS is a generic instrument for the assessment of pain, consisting of a single question that asks participants to record their daily average pain on an 11-point scale, where 0 anchors "no pain" and 10 "pain as bad as you can imagine.
Time Frame: Baseline and EOT (Up to week 8)
Population: FAS population with last observation carried forward (LOCF) imputation.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | ASP0819 15 mg
Number analyzed (Participants) | 94 | 90
Percentage of participants | 30.9 [23.0 to 39.6] | 37.8 [29.2 to 47.0]
Statistical Analysis 1: Comparison: Placebo vs ASP0819 15 mg; Test type: Superiority; p = 0.202, Fisher Exact; [statistical method as in outcome 7, analysis 1]; Difference = 6.9, 90% CI 2-sided [-5.2 to 19.1]

9. Secondary Outcome: Percentage of Participants Achieving ≥ 50 % Reduction From Baseline to Week 8 in Mean Daily Average Pain Score Assessed by NRS
Description: as for outcome 7
Time Frame: Baseline and week 8
Population: FAS with population with BOCF imputation.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | ASP0819 15 mg
Number analyzed (Participants) | 94 | 90
Percentage of participants | 13.8 [8.4 to 21.1] | 15.6 [9.7 to 23.2]
Statistical Analysis 1: Comparison: Placebo vs ASP0819 15 mg; Test type: Superiority; p = 0.451, Fisher Exact; [statistical method as in outcome 7, analysis 1]; Difference = 1.7, 90% CI 2-sided [-10.5 to 13.8]

10. Secondary Outcome: Percentage of Participants Achieving ≥ 50 % Reduction From Baseline to EOT in Mean Daily Average Pain Score Assessed by NRS
Description: as for outcome 7
Time Frame: Baseline and EOT (Up to week 8)
Population: FAS population with LOCF Imputation
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | ASP0819 15 mg
Number analyzed (Participants) | 94 | 90
Percentage of participants | 12.8 [7.5 to 19.9] | 18.9 [12.4 to 27.0]
Statistical Analysis 1: Comparison: Placebo vs ASP0819 15 mg; Test type: Superiority; p = 0.174, Fisher Exact; [statistical method as in outcome 7, analysis 1]; Difference = 6.1, 90% CI 2-sided [-6.2 to 18.1]

11. Secondary Outcome: Change From Baseline in the Fibromyalgia Impact Questionnaire Revised (FIQR) FIQR Function, Symptoms, and Overall Impact Subscales
Description: The 21-item FIQR contains 3 domains: activities of daily living, overall impact, and symptoms. Participants answer each question on an 11-point NRS, with anchors appropriate to each question. The range of function subscale scores will be 0 to 90, with a lower score indicting better (higher) function. The range of overall impact subscale scores will be 0 to 20, with a lower score indicating better (lower) impact. The range of symptoms subscale scores will be 0 to 100, with a lower score indicating a better (lower) level of symptoms. A negative change indicates a reduction/improvement from baseline (i.e. a favorable outcome).
Time Frame: Baseline and weeks 2, 4, 8
Population: FAS population with available data at specified time point.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | ASP0819 15 mg
Number analyzed (Participants) | 94 | 90
Units on a scale
  Week 2: Function Subscale:: number analyzed (Participants) | 90 | 90
  Week 2: Function Subscale: | -8.48 (1.47) | -9.97 (1.46)
  Week 4: Function Subscale: number analyzed (Participants) | 84 | 83
  Week 4: Function Subscale | -9.11 (1.67) | -12.08 (1.66)
  Week 8: Function Subscale: number analyzed (Participants) | 81 | 73
  Week 8: Function Subscale | -11.45 (1.79) | -14.04 (1.82)
  Week 2: Symptom Subscale: number analyzed (Participants) | 90 | 90
  Week 2: Symptom Subscale | -9.20 (1.35) | -10.54 (1.34)
  Week 4: Symptom Subscale: number analyzed (Participants) | 84 | 83
  Week 4: Symptom Subscale | -10.05 (1.51) | -13.78 (1.50)
  Week 8: Symptom Subscale: number analyzed (Participants) | 81 | 73
  Week 8: Symptom Subscale | -11.14 (1.65) | -14.20 (1.68)
  Week 2: Overall Impact Subscale: number analyzed (Participants) | 90 | 90
  Week 2: Overall Impact Subscale | -2.94 (0.45) | -3.94 (0.45)
  Week 4: Overall Impact Subscale: number analyzed (Participants) | 84 | 83
  Week 4: Overall Impact Subscale | -2.95 (0.45) | -4.29 (0.45)
  Week 8: Overall Impact Subscale: number analyzed (Participants) | 81 | 73
  Week 8: Overall Impact Subscale | -3.80 (0.49) | -4.66 (0.49)
Statistical Analysis 1: Comparison: Placebo vs ASP0819 15 mg; Function Subscale: Week 2; Test type: Superiority; p = 0.235, MMRM — MMRM analysis model is performed with change from baseline (Weeks 2, 4, and 8) as response; treatment, center (pooled where necessary), time (Weeks 2, 4 and 8), treatment*time as fixed effects, baseline and baseline*time as covariates; Least Square (LS) Mean difference = -1.48, 90% CI 2-sided [-4.86 to 1.90], Standard Error of Mean 2.04
Statistical Analysis 2: Comparison: Placebo vs ASP0819 15 mg; Function Subscale: Week 4; Test type: Superiority; p = 0.103, MMRM — [p-value comment as in outcome 11, analysis 1]; LSMean Difference = -2.97, 90% CI 2-sided [-6.84 to 0.89], Standard Error of Mean 2.34
Statistical Analysis 3: Comparison: Placebo vs ASP0819 15 mg; Function Subscale: Week 8; Test type: Superiority; p = 0.154, MMRM — [p-value comment as in outcome 11, analysis 1]; LSMean Difference = -2.59, 90% CI 2-sided [-6.78 to 1.60], Standard Error of Mean 2.53
Statistical Analysis 4: Comparison: Placebo vs ASP0819 15 mg; Symptoms Subscale: Week 2; Test type: Superiority; p = 0.238, MMRM — [p-value comment as in outcome 11, analysis 1]; LSMean Difference = -1.34, 90% CI 2-sided [-4.45 to 1.77], Standard Error of Mean 1.88
Statistical Analysis 5: Comparison: Placebo vs ASP0819 15 mg; Symptoms Subscale: Week 4; Test type: Superiority; p = 0.039, MMRM — [p-value comment as in outcome 11, analysis 1]; LSMean Difference = -3.73, 90% CI 2-sided [-7.22 to -0.24], Standard Error of Mean 2.11
Statistical Analysis 6: Comparison: Placebo vs ASP0819 15 mg; Symptoms Subscale: Week 8; Test type: Superiority; p = 0.097, MMRM — [p-value comment as in outcome 11, analysis 1]; LSMean Difference = -3.06, 90% CI 2-sided [-6.93 to 0.81], Standard Error of Mean 2.34
Statistical Analysis 7: Comparison: Placebo vs ASP0819 15 mg; Overall Impact Subscale: Week 2; Test type: Superiority; p = 0.057, MMRM — [p-value comment as in outcome 11, analysis 1]; LSMean DIfference = -0.99, 90% CI 2-sided [-2.03 to 0.04], Standard Error of Mean 0.63
Statistical Analysis 8: Comparison: Placebo vs ASP0819 15 mg; Overall Impact Subscale: Week 4; Test type: Superiority; p = 0.018, MMRM — [p-value comment as in outcome 11, analysis 1]; LSMean Difference = -1.34, 90% CI 2-sided [-2.39 to -0.29], Standard Error of Mean 0.63
Statistical Analysis 9: Comparison: Placebo vs ASP0819 15 mg; Overall Impact Subscale: Week 8; Test type: Superiority; p = 0.111, MMRM — [p-value comment as in outcome 11, analysis 1]; LSMean Difference = -0.86, 90% CI 2-sided [-2.02 to 0.30], Standard Error of Mean 0.70

12. Secondary Outcome: Change From Baseline in the Fibromyalgia Impact Questionnaire Revised (FIQR) FIQR Function, Symptoms, and Overall Impact Subscales
Description: as for outcome 11
Time Frame: Baseline and EOT (Up to week 8)
Population: FAS population with LOCF Imputation.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | ASP0819 15 mg
Number analyzed (Participants) | 94 | 90
Units on a scale
  Function Subscale: EOT | -10.41 (1.66) | -13.55 (1.70)
  Symptom Subscale: EOT | -10.79 (1.52) | -14.07 (1.56)
  Overall Impact Subscale: EOT | -3.40 (0.46) | -4.48 (0.47)
Statistical Analysis 1: Comparison: Placebo vs ASP0819 15 mg; Function Subscale; Test type: Superiority; p = 0.092, ANCOVA — ANCOVA model is performed with change from baseline at the EOT timepoint as response treatment and center (pooled where necessary) as fixed effects and baseline as a covariate; LSMean difference = -3.15, 90% CI 2-sided [-7.05 to 0.75], Standard Error of Mean 2.36
Statistical Analysis 2: Comparison: Placebo vs ASP0819 15 mg; Symptoms subscale; Test type: Superiority; p = 0.065, ANCOVA — [p-value comment as in outcome 12, analysis 1]; LSMean difference = -3.29, 90% CI 2-sided [-6.85 to 0.28], Standard Error of Mean 2.16
Statistical Analysis 3: Comparison: Placebo vs ASP0819 15 mg; Overall Impact Subscale; Test type: Superiority; p = 0.049, ANCOVA — [p-value comment as in outcome 12, analysis 1]; LSMean difference = -1.08, 90% CI 2-sided [-2.15 to -0.01], Standard Error of Mean 0.65

13. Secondary Outcome: Percentage of Participants With Overall Participant Improvement Assessed by Patient Global Impression of Change (PGIC)
Description: The PGIC is a self-administered 7-point Likert scale that asks participants to evaluate their fibromyalgia relative to baseline. PGIC score ranges from 1 to 7, where 1 anchors "Very Much Improved" and 7 anchors "Very Much Worse".
Time Frame: Weeks 2, 4, and EOT (Up to week 8)
Population: FAS population with LOCF imputation.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | ASP0819 15 mg
Number analyzed (Participants) | 94 | 90
Percentage of participants
  Week 2: Very much improved | 3.2 | 2.2
  Week 2: Much Improved | 9.6 | 12.2
  Week 2: Minimally Improved | 31.9 | 42.2
  Week 2: No Change | 44.7 | 34.4
  Week 2: Minimally Worse | 7.4 | 3.3
  Week 2: Much Worse | 2.1 | 4.4
  Week 2: Very Much Worse | 1.1 | 1.1
  Week 4: Very much improved | 3.2 | 4.4
  Week 4: Much Improved | 14.9 | 20.0
  Week 4: Minimally Improved | 31.9 | 28.9
  Week 4: No Change | 33.0 | 37.8
  Week 4: Minimally Worse | 13.8 | 3.3
  Week 4: Much Worse | 3.2 | 4.4
  Week 4: Very Much Worse | 0 | 1.1
  Week EOT: Very much improved | 6.4 | 10.0
  Week EOT: Much Improved | 18.1 | 21.1
  Week EOT: Minimally Improved | 26.6 | 21.1
  Week EOT: No Change | 38.3 | 40.0
  Week EOT: Minimally Worse | 8.5 | 3.3
  Week EOT: Much Worse | 2.1 | 3.3
  Week EOT: Very Much Worse | 0 | 1.1
Statistical Analysis 1: Comparison: Placebo vs ASP0819 15 mg; Week 2; Test type: Superiority — The 90% 2-sided CI is based on profile likelihood and 2-sided p-value is based on likelihood test. p-value is for the comparison of ASP0819 15 mg with Placebo from the above described proportional odds model; p = 0.192, Likelihood test; Odds Ratio (OR) = 1.43, 90% CI 2-sided [0.91 to 2.24]
Statistical Analysis 2: Comparison: Placebo vs ASP0819 15 mg; Week 4; Test type: Superiority; p = 0.285, Likelihod test — The 90% 2-sided CI is based on profile likelihood and 2-sided p-value is based on likelihood test. p-value is for the comparison of ASP0819 15 mg with Placebo from the above described proportional odds model; Odds Ratio (OR) = 1.33, 90% CI 2-sided [0.86 to 2.07]
Statistical Analysis 3: Comparison: Placebo vs ASP0819 15 mg; EOT; Test type: Superiority; p = 0.486, Likelihood test — [p-value comment as in outcome 13, analysis 2]; Odds Ratio (OR) = 1.20, 90% CI 2-sided [0.78 to 1.87]

14. Secondary Outcome: Percentage of Participants With Overall Participant Improvement Assessed by Patient Global Impression of Change (PGIC)
Description: as for outcome 13
Time Frame: Week 8
Population: FAS population with modified last observation carried forward (mLOCF) imputation.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | ASP0819 15 mg
Number analyzed (Participants) | 94 | 90
Percentage of participants
  Week 8: Very much improved | 6.4 | 10.0
  Week 8: Much Improved | 18.1 | 21.1
  Week 8: Minimally Improved | 24.5 | 21.1
  Week 8: No Change | 40.4 | 42.2
  Week 8: Minimally Worse | 8.5 | 3.3
  Week 8: Much Worse | 2.1 | 2.2
  Week 8: Very Much Worse | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs ASP0819 15 mg; Week 8; Test type: Superiority — The 90% 2-sided CI is based on profile likelihood and 2-sided p-value is based on likelihood test; p = 0.305, Likelihood test; Odds Ratio (OR) = 1.32, 90% CI 2-sided [0.85 to 2.05]

ADVERSE EVENTS:
Time Frame: From first dose of study drug until end of study (up to Day 85)
Groups:
- ASP0819: A single oral dose to be taken preferably in the morning with or without food
Arm/Group | Placebo | ASP0819
All-Cause Mortality (participants affected / at risk) | 0/94 | 0/90
Serious Adverse Events (participants affected / at risk) | 0/94 | 0/90
Other Adverse Events (participants affected / at risk) | 27/94 | 30/90
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=94) | ASP0819 (N=90)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 5 (5)
Viral upper respiratory tract infection (Infections and infestations) | 5 (5) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5)
Headache (Nervous system disorders) | 11 (11) | 12 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2016-12-19): https://cdn.clinicaltrials.gov/large-docs/90/NCT03056690/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/90/NCT03056690/SAP_001.pdf